CLINICAL TRIAL: NCT06495645
Title: Computer-aided Gastric Lesion Localization and Miss Rate of Gastric Neoplasms: a Tandem, Randomized Controlled Study
Brief Title: Miss Rate of Gastric Neoplasms Under Computer-aided Endoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lui Ka-Luen, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: protocol_upper_RCTV10
Record Dates: First submitted 2024-06-25; First posted 2024-07-11 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Gastric Neoplasm; Artificial Intelligence
Keywords: Gastric Neoplasm; Artificial intelligence; Miss rate
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-HD group (Experimental): AI-assisted upper gastrointestinal endoscopy follow immediately by high definition (HD) upper gastrointestinal endoscopy
  Interventions: Device: AI-assisted upper gastrointestinal endoscopy
- HD-AI group (Active Comparator): HD upper gastrointestinal endoscopy follow immediately by AI-assisted upper gastrointestinal endoscopy
  Interventions: Device: AI-assisted upper gastrointestinal endoscopy

INTERVENTIONS:
Device: AI-assisted upper gastrointestinal endoscopy — AI-assisted upper gastrointestinal endoscopy

SUMMARY:
This prospective randomized trial compares AI-assisted upper gastrointestinal endoscopy with high definition upper gastrointestinal endoscopy in term of missed rate of gastric neoplasm. The investigators hypothesize the miss rate of high definition upper gastrointestinal endoscopy is higher than AI-assisted upper gastrointestinal endoscopy.

DETAILED DESCRIPTION:
Patients will be randomly assigned to begin with AI-assisted upper gastrointestinal endoscopy follow immediately by high definition (HD) upper gastrointestinal endoscopy (AI-HD group); or start with HD upper gastrointestinal endoscopy follow immediately by AI-assisted upper gastrointestinal endoscopy (HD-AI group). The random allocation sequence is generated by a computer-generated random numerical series, with 1 representing the AI-HD group and 0 representing the HD-AI group. Randomization is conducted in blocks of four at a 1:1 ratio stratified by indications (screening/surveillance vs others), endoscopist's experience (experienced versus less experienced) and mode of sedation (unsedated vs sedated). Experienced endoscopist is defined as qualified endoscopists with more than 7 years experience in upper endoscopy, whereas less experienced endoscopists include fellows and trainees. A research assistant, not directly involved in this study, maintained all randomization codes which are contained within individual opaque envelopes. Upon obtaining patient consent, the envelope will be opened to reveal the assigned examination sequence. Patients remain blinded to their group allocation throughout the study, but the performing endoscopist is aware of the assigned allocation.

Participating endoscopists will receive training on the interpretation of real-time AI detection system as well as detection of dysplasia under HD endoscopy before performing study. All patients will fast for at least 6 hours before the procedure. All examinations will be performed with HD endoscopes (ELUXEO 7000 video system, Fujifilm Co, Tokyo, Japan) under white light. The artificial intelligence assisted gastric dysplasia localization system uses a graphical user interface for real-time display of lesion detection with bounding boxes (Fujifilm Co, Tokyo, Japan).

Each eligible patient will undergo a same-day tandem upper gastrointestinal endoscopy performed by the same endoscopist to evaluate the miss rate of gastric neoplasm. Patients first receive either AI-assisted or HD upper gastrointestinal endoscopy under white light endoscopy, immediately followed by cross-over to other procedure. Endoscopists will be assisted by a research assistant (RS), who activates or deactivates the lesion detection function of AI system between the two examinations. Both first and second examinations are conducted in accordance with the systematic gastric screening protocol, and only the gastric cavity was rescanned during the second observation. The minimal inspection time of the stomach should be 3 minute for the both examination.

Biopsies of all targeted lesions will be taken at the end of each examination. Endoscopists are instructed to biopsy lesions meeting the following criteria in HD examinations: color differences, loss of vascularity, slight elevation or depression, nodularity, thickening, abnormal convergence or flattening of folds, irregular margins, irregular discoloration, or irregular surface. During AI-assisted examinations, targeted lesions are defined as focal lesions marked in localization boxes. Endoscopists are instructed to biopsy areas stably marked with localization boxes that persisted for 5 seconds by the AI system.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40 or older
* Scheduled for elective upper endoscopy

Exclusion Criteria:

* Pregnant women,
* Inability to provide written informed consent
* Prior gastrectomy, and
* Patients deemed unsuitable or high-risk for endoscopy with severe comorbid illnesses

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Gastric neoplasia miss rate | during the intervention
  the number of newly detected gastric neoplasia in the second examination divided by the total number of gastric neoplasia detected in both examinations for each patient.

SECONDARY OUTCOMES:
Gastric neoplasia detection rate | during the intervention
  The proportion of patients with one or more gastric neoplasms detected in the first examination
The biopsy rate | during the intervention
  The proportion of patients who had a biopsy sample taken as a result of the first examination
The number of gastric neoplasms per patient | during the intervention
  The total number of gastric neoplasms detected in the first examination divided by the total number of patients
The miss rate of patients with gastric neoplasms | during the intervention
  The number of patients with a newly detected gastric neoplasm in the second examination divided by the total number of patients with gastric neoplasms detected in both examinations
The positive predictive value (PPV) for gastric neoplasms | during the intervention
  The number of detected gastric neoplasms divided by the number of all targeted lesions in the first examination
Inspection time | during the intervention
  The procedure time of the examinations minus the time taken to obtain a biopsy sample, measured from the passage of the endoscope through the gastroesophageal junction until the completion of the whole examination of the gastric cavity, excluding the inspection time of the duodenum and the biopsy time
The macroscopic and histological types of detected and missed neoplasia in the first examination | during the intervention
  The macroscopic and histological types of detected and missed neoplasia in the first examination
Number of biopsy per patient in the first arm | during the intervention
  Number of biopsy per patient in the first arm
Percentage of positive biopsy | during the intervention
  The number of gastric neoplasm detected divided by total number of biopsy in the first arm

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ka-Luen Lui, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, the University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No